CLINICAL TRIAL: NCT02049177
Title: Alcohol Related Cancers and Genetic Susceptibility in Europe Follow-up - North-West England
Brief Title: Investigation of the Role of Human Papilloma Virus (HPV) in the Prognosis of Head and Neck Cancer
Acronym: ARCAGE-NWE
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: 2/084/13
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Head and Neck Cancer
Keywords: Cancer; Epidemiology; Head and Neck; HPV
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head and Neck Cancer Cases: Cases of Head and Neck Cancer identified in North West England in 2002/2003. Observational study - no intervention other than usual care.

SUMMARY:
Human papilloma virus (HPV) is a recognised cause of some head and neck cancers. Important questions remain however, regarding the role of specific types of HPV, their effect on prognosis and different subtypes of oral, pharyngeal and laryngeal cancer, interaction with other risk factors (such as smoking and alcohol), and potential geographical differences in the effect of HPV.

Via the Alcohol-Related Cancers and Genetic Susceptibility in Europe (ARCAGE) study, which is an international collaboartive case-control study conducted in 15 centres in 11 European countries, and pooling our results with the HPV-AHEAD consortium, we will conduct a systematic analysis of HPV subtypes known or suspected to be involved in head and neck cancer. This will involve investigation of HPV risk by tumour site (oral, oropharynx, hypopharynx, larynx), tumour stage, country, sex and age, and whether risk is modified by exposure to other known or suspected carcinogens including tobacco, alcohol and medical history.

It is intended that this work will contribute to the development of evidence that may feed into treatment protocols for these cancers as well as evaluations of the feasibility for extending HPV vaccine programs.

ELIGIBILITY:
Inclusion Criteria:

* Consent to follow-up and use of tissue samples

Exclusion Criteria:

* No existing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases that were previously identified for the HPV-AHEAD case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
HPV type | From surgical/biopsy samples taken in 2002/2003, to be typed in 2014

SECONDARY OUTCOMES:
Vital status | 2014
Cancer Reccurrence | 2002-2014
Secondary cancers | 2002-2014

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn
  - Blackpool Victoria Infirmary, Blackpool
  - Manchester Royal Infirmary, Manchester
  - North Manchester General Hospital, Manchester
  - The Christie Hospital, Manchester
  - Royal Preston Hospital, Preston

REFERENCES:
- See also: Study Website — http://arcage.iarc.fr/